CLINICAL TRIAL: NCT01533701
Title: Biosampling for Markers of Hypoxia in Fetal Blood Scalp Sampling During Labor
Brief Title: Scalp Sampling for Fetal Surveillance
Acronym: FBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Maria Jonsson, Principal investigator, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UASKK2012
Record Dates: First submitted 2012-02-06; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Fetal Hypoxia
Keywords: Hypoxia; Fetal blood sampling; Lactate; pH; base deficit; angiogenic factors; suspected fetal hypoxia
MeSH Terms: conditions — Fetal Hypoxia; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fetal scalp blood scalp, amniotic fluid, maternal blood and umbilical cord sampling — Fetal blood sampling is conducted when a non reassuring cardiotocographic pattern occurs to detect fetal hypoxia during labor. Amniotic fluid, maternal blood is sampled in cases of fetal blood sampling. Umbilical cord blood sampling is conducted at delivery.

SUMMARY:
The purpose of this study is to compare lactate and total acid-base status in fetal scalp blood with lactate and total acid-base status in maternal blood and amniotic fluids to provide information on how lactate and base deficit correlates with scalp samples.

Furthermore, the investigators want to study whether angiogenic factors in fluids above may be a possible marker of asphyxia during labor.

ELIGIBILITY:
Inclusion Criteria:

* All deliveries eligible for fetal blood sampling

Exclusion Criteria:

* Non Swedish speaking
* Those who decline to participate in the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Hypoxia | 120 seconds
  Fetal blood sampling is conducted when a non reassurring cardiotocographic pattern occurs to detect fetal hypoxia during labor

SECONDARY OUTCOMES:
Subacute hypoxia | 120 seconds
  Fetal blood sampling is conducted when a non reasurring cardiotocographic pattern occurs to detect fetal hypoxia during labor

CONTACTS AND LOCATIONS:
Locations (1):
- Delivery department Uppsala University hospital, Uppsala, Sweden